CLINICAL TRIAL: NCT07390110
Title: Comparative Effectiveness of Oral Semaglutide vs Sitagliptin Among Individuals With Heart Failure With Preserved Ejection Fraction (STEP-HFpEF DM ORAL)
Status: Active, not recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor, Brigham and Women's Hospital
Other Study IDs: 2018P002966-STEP-HFpEF DM ORAL
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes; Heart Failure
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure | interventions — semaglutide; Sitagliptin Phosphate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Initiation of oral semaglutide: Exposure group: Semaglutide in the oral formulation in any dose.
  Interventions: Drug: Oral semaglutide
- Initiation of sitagliptin: Reference group: Sitagliptin in the oral formulation in any dose
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Oral semaglutide — Initiation of semaglutide dispensing claim is used as the exposure.
  Groups: Initiation of oral semaglutide
Drug: Sitagliptin — Initiation of sitagliptin dispensing claim is used as the reference.
  Groups: Initiation of sitagliptin

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale emulation of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the Randomized Controlled Trials Duplicated Using Prospective Longitudinal Insurance Claims: Applying Techniques of Epidemiology (RCT-DUPLICATE) initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to assess the comparative effectiveness of oral semaglutide vs sitagliptin as a placebo proxy using a target trial emulation framework. The SOUL trial (NCT03914326) and its database emulation study (NCT06659718) demonstrated a reduction in atherosclerotic cardiovascular events with oral semaglutide among patients with type 2 diabetes and high cardiovascular risk. The STEP-HF-EF DM trial (NCT04916470) and its database emulation study (NCT06914102) found the injectable formulation of semaglutide to lower the risk for heart failure hospitalization in patients with cardiometabolic HFpEF, and its non-inferiority to tirzepatide (NCT06914141). However, the effectiveness of oral semaglutide in reducing the risk of heart failure events remains unclear.

The comparative effectiveness target trial described below draws from eligibility criteria from the STEP-HFpEF DM trial but is designed to include a much larger and more diverse group of patients than the trial allowed. Although many features of the target trial cannot be directly replicated in healthcare claims, measurements of key design features, including outcomes, exposures, and inclusion/exclusion criteria, were designed to proxy those features from the target trial. Randomization cannot be achieved in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice.

The database study will be a new-user active-comparative study, conducted using 3 national United States claims databases, where we compare the effect of oral semaglutide vs sitagliptin on heart failure outcomes.

ELIGIBILITY:
Eligible Cohort Entry Dates:

* Optum: Eligible cohort entry period from September 20, 2019 to November 30, 2025.
* Marketscan: Eligible cohort entry from September 20, 2019 to December 31, 2023.
* Medicare: Eligible cohort entry from September 20, 2019 to December 31, 2020.

Inclusion Criteria:

* Heart failure
* BMI > 27.0kg/m2
* Type 2 diabetes mellitus
* LVEF > 45%
* Age > 18 years
* Sex: male or female

Exclusion Criteria:

* Multiple endocrine neoplasia type 2 or medullary thyroid carcinoma, other malignancy
* Type 1 diabetes mellitus, uncontrolled diabetic retinopathy or maculopathy, bariatric surgery, end-stage renal disease or dialysis, nursing home admission
* Any use of GLP-1-RA including injectable semaglutide except oral semaglutide, pregnancy, treatment with continuous subcutaneous insulin infusion
* Concurrent use of both study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals aged 18 years or older with heart failure with preserved ejection fraction.
Sampling Method: Non-Probability Sample
Enrollment: 25664 (Actual)
Dates: Start 2026-01-24 (Actual); Primary Completion 2026-02-11 (Estimated); Study Completion 2026-02-11 (Estimated)

PRIMARY OUTCOMES:
Composite of worsening heart failure event (exacerbated symptoms of heart failure resulting in hospitalization, intravenous diuretic therapy in an urgent care setting) or all-cause mortality. | Through study completion until the first of outcome, disenrollment, end of study period, discontinuation (45 days grace and risk window), switch between the arms, start of any other GLP-1-RA including injectable semaglutide.
  To evaluate the comparative effect of oral semaglutide vs sitagliptin on the composite of worsening heart failure events or all-cause mortality in patients with heart failure with preserved ejection fraction in clinical practice.
Worsening heart failure event (exacerbated symptoms of heart failure resulting in hospitalization, intravenous diuretic therapy in an urgent care setting). | Through study completion until the first of outcome, disenrollment, end of study period, discontinuation (45 days grace and risk window), switch between the arms, start of any other GLP-1-RA including injectable semaglutide.
  To evaluate the comparative effect of oral semaglutide vs sitagliptin on worsening heart failure events with heart failure with preserved ejection fraction in clinical practice.

SECONDARY OUTCOMES:
Heart failure hospitalization. | Through study completion until the first of outcome, disenrollment, end of study period, discontinuation (45 days grace and risk window), switch between the arms, start of any other GLP-1-RA including injectable semaglutide.
  To evaluate the comparative effect of oral semaglutide vs sitagliptin on heart failure hospitalization in patients with heart failure with preserved ejection fraction in clinical practice.
Worsening heart failure event requiring intravenous diuretic therapy in an urgent care setting. | Through study completion until the first of outcome, disenrollment, end of study period, discontinuation (45 days grace and risk window), switch between the arms, start of any other GLP-1-RA including injectable semaglutide.
  To evaluate the comparative effect of oral semaglutide vs sitagliptin on worsening heart failure events in patients with heart failure with preserved ejection fraction in clinical practice.
Urinary tract infections. | Through study completion until the first of outcome, disenrollment, end of study period, discontinuation (45 days grace and risk window), switch between the arms, start of any other GLP-1-RA including injectable semaglutide.
  To evaluate the comparative effect of oral semaglutide vs sitagliptin on the safety outcome of urinary tract infections in clinical practice.
Serious infections. | Through study completion until the first of outcome, disenrollment, end of study period, discontinuation (45 days grace and risk window), switch between the arms, start of any other GLP-1-RA including injectable semaglutide.
  To evaluate the comparative effect of oral semaglutide vs sitagliptin on the safety outcome of serious infections in clinical practice.
Gastrointestinal adverse events. | Through study completion until the first of outcome, disenrollment, end of study period, discontinuation (45 days grace and risk window), switch between the arms, start of any other GLP-1-RA including injectable semaglutide.
  To evaluate the comparative effect of Oral semaglutide vs sitagliptin on the safety outcome of gastrointestinal adverse events in clinical practice.

OTHER OUTCOMES:
Hernia (excluding patients with recent outcome prior to the follow-up time window (30 days)). | Through study completion until the first of outcome, disenrollment, end of study period, discontinuation (45 days grace and risk window), switch between the arms, start of any other GLP-1-RA including injectable semaglutide.
  To evaluate the effect of oral semaglutide vs sitagliptin on a negative control outcome of hernia in clinical practice.
Lumbar radiculopathy (excluding patients with recent outcome prior to the follow-up time window (30 days)). | Through study completion until the first of outcome, disenrollment, end of study period, discontinuation (45 days grace and risk window), switch between the arms, start of any other GLP-1-RA including injectable semaglutide.
  To evaluate the effect of oral semaglutide vs sitagliptin on a negative control outcome of lumbar radiculopathy in clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital; Nils Krüger, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol (2026-01-24): https://cdn.clinicaltrials.gov/large-docs/10/NCT07390110/Prot_000.pdf